CLINICAL TRIAL: NCT01342107
Title: The Effect of Alcon Multi-Purpose Disinfecting Solution (MPDS) on Lens Wettability
Brief Title: Effect of FID 114675A on Lens Wettability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: C-10-024
Record Dates: First submitted 2011-01-07; First posted 2011-04-27 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Contact Lens Wettability
Keywords: Contact Lenses; Contact Lens Care; Multi-Purpose Solution Wettability; Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114675A (Experimental): Contact lens soaked overnight in an investigational multi-purpose disinfecting solution randomly assigned to one eye, with contact lens removed directly from the blister pack assigned to the fellow eye for contralateral wear. Both products worn for one day, 16 hours.
  Interventions: Device: FID 114675A multi-purpose disinfecting solution (MPDS); Device: Soft contact lens
- Blister Pack (Active Comparator): Contact lens removed directly from the blister pack randomly assigned to one eye, with contact lens soaked overnight in an investigational multi-purpose disinfecting solution assigned to the fellow eye for contralateral wear. Both products worn for one day, 16 hours.
  Interventions: Device: Soft contact lens; Device: Blister pack solution

INTERVENTIONS:
Device: FID 114675A multi-purpose disinfecting solution (MPDS) — Investigational multi-purpose disinfecting solution intended for use as a cleaning, reconditioning, rinsing, disinfecting, and storage solution for silicone hydrogel and soft contact lenses.
  Arms: FID 114675A
Device: Soft contact lens — Soft hydrogel or silicone hydrogel contact lens matching subject's pre-study lens, including parameters, worn 16 hours on day of dispense.
  Other Names: Acuvue2; PureVision; Acuvue Oasys
Device: Blister pack solution — Commercially approved storage solution as found in the contact lens blister pack.
  Other Names: Acuvue2; PureVision; Acuvue Oasys
  Arms: Blister Pack

SUMMARY:
The purpose of this study is to evaluate lens wettability of contact lenses when used with an investigational multi-purpose disinfecting solution.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or age or older with normal eyes, other than correction for refractive error.
* At least 5 days successful daily wear (minimum 8 hours per day) of PureVision®, Acuvue® Oasys™, or Acuvue® 2 contact lenses prior to Visit 1
* Vision correctable to 20/30 (Snellen) or better in each eye at distance with lenses at Visit 1 (Day 0 - Baseline).
* Grade 0 or Grade 1 wettability in both eyes after at least 15 minutes of lens wear at Visit 1 (Day 0 - Baseline).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the test articles or affect the results of the study.
* Need to wear contact lenses on an extended wear basis (i.e., overnight) during the study.
* Use of products other than a multi-purpose solution or hydrogen peroxide solution, including daily and enzyme cleaners and saline rinses, for lens care at least 7 days prior to Visit 1 (Day 0 - Baseline).
* Use of over-the-counter (OTC) or prescribed topical ocular medications within 7 days prior to Visit 1. Use of lens rewetting drops is acceptable.
* History or current ocular infections or ocular inflammatory events.
* Ocular surgery within the past year.
* Participation in any investigational study within the past 30 days.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FID 114675A: Contact lens soaked overnight in an investigational multi-purpose disinfecting solution randomly assigned to right eye, with contact lens removed directly from the blister pack assigned to left eye for contralateral wear.
- Blister Pack: Contact lens removed directly from the blister pack randomly assigned to right eye, with contact lens soaked overnight in an investigational multi-purpose disinfecting solution assigned to left eye for contralateral wear.
Period: Overall Study
Arm/Group | FID 114675A | Blister Pack
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FID 114675A | Blister Pack | Total
Number analyzed (Participants) | 34 | 32 | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 36.6 (10.76) | 37.3 (12.34) | 36.9 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Lens Wettability
Description: As assessed by the investigator during slit-lamp exam and rated on a 0-4 scale, with 0 = a smooth uniformly reflecting wettable surface; 1 = a coarse hazy wettable surface which seems resolved momentarily with each blink and becomes exacerbated with staring; 2 = one stable dry (non-wetting) area of some magnitude; 3 = more than one stable dry (non-wetting) area of some magnitude; 4 = non-wettable lens surface of severe magnitude. Lenses with a Grade 0 or 1 were rated as wettable and reported as a percentage of total lenses evaluated.
Time Frame: 16 hours
Population: Intent to treat. All subject-eyes that received contact lenses pre-soaked per treatment regimen and completed Visit 2 (Day 1 - Exit at 16 hours) were included in the ITT data set.
Measure: Number (95% Confidence Interval); unit: percentage of lenses
Groups:
- FID 114675A: Contact lens soaked overnight in an investigational multi-purpose disinfecting solution and inserted on day of dispense for 16 hours of wear.
- Blister Pack: Contact lens removed directly from the blister pack and inserted on day of dispense for 16 hours of wear.
Arm/Group | FID 114675A | Blister Pack
Number analyzed (Participants) | 66 | 66
percentage of lenses | 95.5 [87.3 to 99.1] | 97.0 [89.5 to 99.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: October 11, 2010 through February 2, 2011.
Description: All subjects who received contact lenses pre-soaked per treatment regimen were evaluable for the safety analysis.
Arm/Group | FID 114675A | Blister Pack
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.